CLINICAL TRIAL: NCT07175350
Title: Valutazione Della "Financial Toxicity" Nei Pazienti Sottoposti a Radioterapia: Uno Studio Multicentrico Italiano Promosso da yAIRO (Associazione Italiana Radioterapia e Ocologia Clinica)
Brief Title: Financial Toxicity (FT) for Radiotherapy (RT) Patients in Italy: a yAIRO (Associazione Italiana Radioterapia e Ocologia Clinica) Multicenter Study
Acronym: FIT-RT
Status: Recruiting | Type: Observational
Sponsor: Valerio Nardone (Other)
Collaborators: National Cancer Institute (NCI), Naples (Unknown)
Responsible Party: Sponsor-Investigator, Valerio Nardone, Clinical Professor, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Other Study IDs: FIT-RT
Record Dates: First submitted 2025-08-01; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Oncologic Diseases
Keywords: Oncologic Diseases; Radiotherapy; Financial toxicity; PROFFIT questionnaire; Quality of Life
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncologic patients undergoing radiotherapy
  Interventions: Other: PROFFIT

INTERVENTIONS:
Other: PROFFIT — The PROFFIT questionnaire is a PRO instrument composed by 16 items encompassing all the major life domains where FT can be expressed and is formed by two type of items: (1) outcome (items 1-7) and (2) determinants (items 8-16); EORTC QLQ-C30 questionnaire is a 30-item questionnaire that measures health-related quality of life (HRQOL) in cancer patients ; PRO-CTCAE is a short list of 43 symptoms relevant for ovarian cancer
  Other Names: EORTC QLQ-C30 questionnaire; PRO-CTCAE

SUMMARY:
Non- profit, multicenter, prospective, observational study. The study aims to assess financial toxicity (FT) in patients undergoing radiotherapy for oncological diseases, assessed with a validated questionnaire (Patient Reported Outcome for Fighting FInancial Toxicity-PROFFIT- questionnaire).

DETAILED DESCRIPTION:
PROFFIT questionnaire is an Italian instrument for evaluating FT in cancer patients in the Italian healthcare context. It includes 16 total items, 7 measuring FT (defining the PROFFIT financial score) and 9 measuring possible determinants of FT. The primary objective of the study is to assess FT in patients undergoing radiotherapy for oncological diseases and compare FT in different patients group defined according to baseline characteristics (oncologic disease, type of radiotherapy and treatment, age and sex).

Primary comparison will be based on PROFFIT questionnaire fulfilled at baseline (before starting radiotherapy), at the end of RT treatment, at first follow-up visit (1-2 months after the end of RT).

Exploratory analyses will be conducted to verify whether changes in the FT score during treatment are correlated with QOL (EORTC QLQ-C30 questionnaire), toxicity (PRO-CTCAE), and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age.

Histological diagnosis of malignancy for which the patient requires radiotherapy treatment.

Exclusion Criteria:

* Patient refusal to complete the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologic patients undergoing radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Financial toxicity (PROFFIT financial score and "determinants") | baseline (before starting RT), periprocedural (end of radiotherapy treatment, average of 1-2 months); 1-2 months after the end of RT(first follow-up visit) up to 12 months.
  PROFFIT financial score is defined according to items 1-7 of the PROFFIT questionnaire. It will be calculated according to published rules (Riva S, et al. BMJ Open. 2019 Sep;9(9):e031485). The baseline score for determinants (items 8-16) and their change during treatment

OTHER OUTCOMES:
Quality of Life (QoL) | baseline (before starting RT), periprocedural (end of radiotherapy treatment, average of 1-2 months); 1-2 months after the end of RT(first follow-up visit) up to 12 months.
  QoL will be assessed using EORTC QLQ-C30 questionnaire and selected symptoms of the PRO-CTCAE library.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Grassi, MD, Principal Investigator — AOU "L. Vanvitelli" - UOC Radioterapia
Locations (7):
- Italy (7):
  - Radioterapia Oncologica - Ospedale Mons. Dimiccoli, Barletta
  - Unità di Radioterapia - Responsible Research Hospital, Campobasso
  - Radioterapia oncologica - Ospedale "Vito Fazzi" -, Lecce
  - AOU "L. Vanvitelli" - UOC Radioterapia, Napoli
  - .C. Radioterapia - INT G. Pascale, Napoli
  - Radioterapia Oncologica, IRCCS-CROB, Potenza
  - UOC Radioterapia - Fondazione Policlinico A. Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Undecided